CLINICAL TRIAL: NCT00095693
Title: Phase II Study of BAY 43-9006 in Patients With Metastatic Thyroid Carcinoma
Brief Title: Sorafenib Tosylate in Treating Patients With Locally Advanced, Metastatic, or Locally Recurrent Thyroid Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01457; NCI-2012-01457 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU-0441; CDR0000393968; NCI-6608; OSU-2004C0068; OSU 0441 (Other: Ohio State University Medical Center); 6608 (Other: CTEP); N01CM62207 (NIH); P30CA016058 (NIH); N01CM62206 (NIH); U01CA076576 (NIH)
Record Dates: First submitted 2004-11-05; First posted 2004-11-08 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Anaplastic Thyroid Cancer; Insular Thyroid Cancer; Recurrent Thyroid Cancer; Stage III Follicular Thyroid Cancer; Stage III Papillary Thyroid Cancer; Stage IV Follicular Thyroid Cancer; Stage IV Papillary Thyroid Cancer
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic; Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary | interventions — Sorafenib; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

ARMS (1):
- Treatment (sorafenib tosylate) (Experimental): Patients receive oral sorafenib tosylate twice daily for up to 6 months in the absence of disease progression or unacceptable toxicity. Patients achieving CR receive 8 additional weeks of therapy beyond CR.
  Interventions: Drug: sorafenib tosylate; Other: laboratory biomarker analysis; Other: pharmacological study; Radiation: fludeoxyglucose F 18; Procedure: positron emission tomography; Procedure: dynamic contrast-enhanced magnetic resonance imaging

INTERVENTIONS:
Drug: sorafenib tosylate — Given PO
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Radiation: fludeoxyglucose F 18 — Correlative studies
  Other Names: 18FDG; FDG
Procedure: positron emission tomography — Correlative studies
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: dynamic contrast-enhanced magnetic resonance imaging — Correlative studies
  Other Names: DCE-MRI

SUMMARY:
Phase II trial to study the effectiveness of sorafenib tosylate in treating patients who have locally advanced, metastatic, or locally recurrent thyroid cancer. Sorafenib tosylate may stop the growth of tumor cells by blocking the enzymes necessary for their growth and by stopping blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine objective response rate in patients with locally advanced, metastatic, or locally recurrent differentiated thyroid cancer treated with sorafenib (BAY 43-9006).

SECONDARY OBJECTIVES:

I. Determine the toxicity of this drug in these patients. II. Correlate thyroglobulin levels with tumor response in patients treated with this drug.

III. Correlate fludeoxyglucose F 18 positron emission tomography results with tumor response in patients treated with this drug.

IV. Correlate tumor permeability and vascularity, as determined by dynamic contrast-enhanced MRI, with tumor response in patients treated with this drug.

V. Determine the pharmacodynamics of this drug in these patients. VI. Correlate the presence and type of B-raf, N-ras, or RET/PTC gene mutations with clinical response in patients treated with this drug.

VII. Correlate the degree of Ras-MAPK signaling inhibition and vascular endothelial growth factor expression with clinical response in patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to diagnosis (papillary thyroid cancer that is chemo-naïve vs all others).

Patients receive oral sorafenib tosylate twice daily for up to 6 months in the absence of disease progression or unacceptable toxicity. Patients achieving complete remission (CR) receive 8 additional weeks of therapy beyond CR.

Patients are followed within 2-4 weeks after completion of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of 1 of the following:

  * Papillary thyroid cancer (stratum I)
  * Papillary, follicular, Hurthle cell, insular, or anaplastic thyroid cancer (stratum II)

    * Mixed histology, poorly differentiated, or tall-cell variants allowed
* Metastatic, locally advanced, or locally recurrent disease
* At least 1 unidimensionally measurable lesion >= 20 mm by conventional techniques OR >= 10 mm by spiral CT scan

  * The following are considered non-measurable disease:

    * Tumors in a previously irradiated area
    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
* Archival tumor tissue block OR material collected before study entry available (stratum I)
* Biopsy-accessible disease (stratum I)
* Performance status - ECOG 0-1
* At least 6 months
* WBC >= 3,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* No bleeding diathesis
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* AST and ALT =< 1.5 times ULN
* Creatinine =< 1.5 times ULN
* No uncontrolled hypertension
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing to undergo 2 tumor biopsies during study participation (stratum I)
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to sorafenib
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No other concurrent malignancy except nonmetastatic nonmelanoma skin cancer or carcinoma in situ of the cervix
* No prior systemic chemotherapy for thyroid cancer (stratum I)

  * Prior systemic chemotherapy used to treat a second primary cancer with curative intent allowed provided the primary cancer was treated more than 5 years before study entry
* No more than 3 prior systemic chemotherapy regimens for thyroid cancer (stratum II)
* More than 6 weeks since prior systemic chemotherapy (stratum II)
* No prior external beam radiotherapy to the sole site of measurable disease (except for patients with anaplastic thyroid cancer)
* More than 6 weeks since prior external beam radiotherapy
* More than 24 weeks since prior iodine I 131
* Recovered from all prior therapy
* No prior sorafenib
* More than 6 weeks since prior investigational tumor-specific therapy
* Concurrent oral or IV bisphosphonates for bony metastases allowed at the discretion of the investigator
* No other concurrent tumor-specific or investigational therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent therapeutic anticoagulation

  * Concurrent prophylactic anticoagulation (e.g., low-dose warfarin) for venous or arterial access devices allowed provided PT, INR, or PTT are normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-10; Primary Completion 2005-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Up to 4 weeks
  The 95% confidence intervals should be provided.

SECONDARY OUTCOMES:
Incidence of toxicity | Up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Shah, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States